CLINICAL TRIAL: NCT02261662
Title: Randomized Controlled Study of Off-Label Use of Ribavirin in Management of Mucocutaneous Extrahepatic Manifestations of HCV Infection
Brief Title: Off-Label Use of Ribavirin in Management of Mucocutaneous Extrahepatic Manifestations of HCV Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Shebl, Dr., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin HCV mucocutaneous
Record Dates: First submitted 2014-09-26; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis C; Lichen Planus; Vasculitis; Autoimmune Diseases
MeSH Terms: conditions — Hepatitis C; Lichen Planus; Vasculitis; Autoimmune Diseases | interventions — Ribavirin; Betamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ribavirin and Betamethasone (Experimental): A nucleoside antimetabolite antiviral agent that blocks nucleic acid synthesis and is used against both RNA and DNA viruses.
  It will be used along with Topical steroids; Betamethasone
  Interventions: Drug: Ribavirin; Drug: Betamethasone
- Betamethasone alone (Experimental): Topical steroids alone will be used; Betamethasone.
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Ribavirin — A nucleoside antimetabolite antiviral agent that blocks nucleic acid synthesis and is used against both RNA and DNA viruses.
  It will be used along with Topical steroids; Betamethasone
  Other Names: Copegus
  Arms: Ribavirin and Betamethasone
Drug: Betamethasone — Topical Steroids alone will be used; Betamethasone
  Other Names: Corticosteroid

SUMMARY:
This study will be conducted on 30 patients with mucocutaneous complaints and documented HCV infection. The study will be done at Tropical medicine department , Tanta university. It will be conducted between June2014 and November 2014.

The aim of the study is to assess efficacy of Ribavirin in the management of mucocutaneous extrahepatic manifestations of HCV infection.

DETAILED DESCRIPTION:
Hepatitis C virus is a common cause of chronic liver disease worldwide and represent public health problem. The Egyptian Demographic Health Survey (EDHS), a cross sectional survey including hepatitis C virus (HCV) biomarkers, was conducted in 2008 on a large nationally representative sample. It estimated HCV prevalence among the 15-59 years age group to be 14.7% . Accordingly, Egypt has the highest HCV prevalence in the world.

Although HCV is a hepatotropic virus, in some patients the primary manifestations of infection occur outside the liver. There is a growing body of evidence to support the idea that HCV can replicate efficiently in extrahepatic tissues including the Peripheral blood mononuclear cells (PBMC). Autoimmune manifestations are common in patients chronically infected by HCV . These manifestations can be dominant, whereas the hepatic disease can be quiescent or mild. More recently, there has been growing interest in the relationship between HCV and Sjogren's syndrome (SS), rheumatoid arthritis (RA), and systemic lupus erythematosus (SLE).

Of those , this article is interested in cutaneous and mucous membrane manifestations where many reports have shown that cutaneous manifestations are often the first signs of chronic HCV infection and these are indicated in 20-40% of the patients presenting to the dermatology clinics, therefore dermatologists must be aware of skin disorders associated with viral infection. The most commonly encountered dermatological manifestations of HCV infection includes mixed cryoglobulinemia (MC), porphyria cutanea tarda (PCT), cutaneous and/or oral lichen planus (LP), urticaria, pruritus, thrombocytopenic purpura and cutaneous vasculitis. Although majority of skin manifestations of chronic HCV infection represent the clinical impression of autoimmune phenomena, however, precise pathogenesis of these extra-hepatic complications is not well understood.

The aim of the study is to assess efficacy of Ribavirin in the management of mucocutaneous extrahepatic manifestations of HCV infection

This study will be conducted on 30 patients with mucocutaneous complaints and documented HCV infection. The study will be done at Tropical medicine department , Tanta university. It will be conducted between June2014 and November 2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of HCV infection and mucocutaneous complaint and contraindicated to have standard antiviral therapy.

Exclusion Criteria:

* Hypersensitivity to Ribavirin
* Pregnant & Lactating women
* Male partners of pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with improved skin manifestations of HCV infection after taking Ribavirin compared with topical steroids. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, MD, Principal Investigator — Tanta Faculty of Medicine, Professor; Fat-heya E Assel, MD, Study Director — Tanta Faculty of Medicine, Professor; Mohamed Y Rabei, Study Director — Dr.; Islam S Ismail, Study Director — Dr.
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Result] Alter MJ. Epidemiology of hepatitis C virus infection. World J Gastroenterol. 2007 May 7;13(17):2436-41. doi: 10.3748/wjg.v13.i17.2436. PMID 17552026
- [Result] Alavian SM. Hepatitis C infection in Iran; A review article. Iran J Clin Infect Dis. 2009;4(1):47-59
- [Result] Kaldor JM, Dore GJ, Correll PK. Public health challenges in hepatitis C virus infection. J Gastroenterol Hepatol. 2000 May;15 Suppl:E83-90. doi: 10.1046/j.1440-1746.2000.02134.x. PMID 10921388
- [Result] Patrick DM, Buxton JA, Bigham M, Mathias RG. Public health and hepatitis C. Can J Public Health. 2000 Jul-Aug;91 Suppl 1:S18-21, S19-23. English, French. PMID 11059125
- [Result] Prati F, Lodi V, D'Elia V, Truffelli D, Lalic H, Raffi GB. Screening of health care workers for hepatitis B virus and hepatitis C virus: criteria for fitness for work. Arh Hig Rada Toksikol. 2000 Mar;51(1):19-26. PMID 11059069
- [Result] Alavian SM, Kabir A, Ahmadi AB, Lankarani KB, Shahbabaie MA, Ahmadzad-Asl M. Hepatitis C infection in hemodialysis patients in Iran: a systematic review. Hemodial Int. 2010 Jul;14(3):253-62. doi: 10.1111/j.1542-4758.2010.00437.x. Epub 2010 May 17. PMID 20491973
- [Result] El-Zanaty F, Way A. Egypt Demographic and Health Survey 2008. Egyptian: Ministry of Health. Cairo: El-Zanaty and Associates and Macro International; 2009. p. 431.
- [Result] Shepard CW, Finelli L, Alter MJ. Global epidemiology of hepatitis C virus infection. Lancet Infect Dis. 2005 Sep;5(9):558-67. doi: 10.1016/S1473-3099(05)70216-4. PMID 16122679
- [Result] Clifford BD, Donahue D, Smith L, Cable E, Luttig B, Manns M, Bonkovsky HL. High prevalence of serological markers of autoimmunity in patients with chronic hepatitis C. Hepatology. 1995 Mar;21(3):613-9. PMID 7533120
- [Result] Galossi A, Guarisco R, Bellis L, Puoti C. Extrahepatic manifestations of chronic HCV infection. J Gastrointestin Liver Dis. 2007 Mar;16(1):65-73. PMID 17410291
- [Result] Poljacki M, Gajinov Z, Ivkov M, Matic M, Golusin Z. [Skin diseases and hepatitis virus C infection]. Med Pregl. 2000 Mar-Apr;53(3-4):141-5. Croatian. PMID 10965678
- [Result] Cordel N, Chosidow O, Frances C. Cutaneous disorders associated with hepatitis C virus infection. Ann Med Interne (Paris). 2000 Feb;151(1):46-52. PMID 10761562